CLINICAL TRIAL: NCT03161444
Title: Estimated Cumulative Incidence of Zika Infection at the End of the First Epidemic in the French West Indies in a Sample of Patients Followed for HIV Infection.
Acronym: ZIKAVIH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Active circulation of dengue virus in the region of the study that may affect the result of zika serology
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: University Hospital of Guadeloupe (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16/B/06; 2016-A01173-48 (Other: ANSM)
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: HIV Infections; Zika Virus Infection
MeSH Terms: conditions — HIV Infections; Zika Virus Infection

STUDY DESIGN:
Intervention Model Description: A blood sample collection for the study will be taken to each participant. Each subject enrolled must have previously participated in the study CHIKVIH.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elective patient (Other): Patient who has patricipated to the study CHIKVIH (NCT02553369) will have a blood collection during a follow up visit for HIV infection.
  Interventions: Other: Biological sample collection

INTERVENTIONS:
Other: Biological sample collection — A blood sample collection for the study will be taken to each participant Each subject enrolled must have previously participated to the study CHIKVIH.

SUMMARY:
This study will estimate the cumulative incidence of Zika infection at the end of the first epidemic in the French West Indies in a sample of patients followed for HIV infection.

DETAILED DESCRIPTION:
Zika virus infection is expanding in all tropical and subtropical areas. The presence of Aedes albopictus in southern France raises concerns about the occurrence of outbreaks of indigenous Zika virus transmission. In this context, knowledge of the cumulative impact of the epidemic that affected the Caribbean in 2016 is an important issue for the management of future epidemics and modeling work. Since the Zika virus has not yet been circulated in the Lesser Antilles, the cumulative incidence rate can be estimated by conducting a general population seroprevalence survey at the end of the epidemic, or more simply within a cohort of patients regularly monitored and whose habitat is distributed throughout the study area. Thus, HIV-infected patients who benefit from regular clinical biological monitoring constitute a population sample perfectly adapted to the study of the emergence of the Zika virus in the French West Indies. The cumulative incidence of infection with the chikungunya virus after the 2014 epidemic has thus been estimated at 58% for Martinique and Guadeloupe using this method.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years pold)
* Followed for HIV infection at the 2 investigators centers (1 located at Martinique and 1 at Guadeloupe)
* Resident in Martinique /Guadeloupe (French West Indies) betwwen 01JAN2016 and 31DEC2016
* Affiliate or beneficiary of a social security scheme.
* Informed consent signed by the patient

Exclusion Criteria:

* Patient who has stayed in another area at risk of transmission of the Zika virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Presence or not of Zika virus-specific immunoglobulin G antibodies in the serum taken after the epidemic | 1 day
  Presence or absence of ZIKV-specific IgG antibodies in the serum taken at the end of the Zika epidemic within six months of the official end of the epidemic for each territory of the French west Indies

SECONDARY OUTCOMES:
Existence or not of clinical signs evocating of an episode of disease with Zika virus. | 1 day during the study
  The clinician in charge of the patient will question him about the occurrence of a clinical episode suggestive of Zika virus infection during the epidemic
Presence or not of Dengue virus specific antibodies before the outbreak of Zika virus infection, sought on the samples taken at the end of the chikungunya epidemic. | 1 day on biological sample collected before the outbreak of Zika virus
  Serological analysis will be performed on biological sample collected in the frame of the heath follow-up of teh patient and stored before the epidemic of Zika Virus disease
Presence or not of Chikungunya-specific antibodies before the outbreak of Zika virus infection, sought after sampling at the end of the chikungunya epidemic. | 1 day on biological sample collected before the outbreak of Zika virus
  Serological analysis will be performed on biological sample collected in the frame of the heath follow-up of teh patient and stored before the epidemic of Zika Virus disease
Evolution of the CD4 lymphocyte levels before and after the outbreak of Zika virus | 6 months before the outbreak of Zika virus ; 12 months of the outbreak of Zika virus; First 6 months after the outbreak of Zika virus
  All biological results for CD4 Lymphocyte will be collected retrospectivelly : 6 months before the outbreak of Zika virus , 12 months of the outbreak of Zika virus and 6 months after the outbreak of Zika virus in order to observe its evolution
Evolution of the HIV1 RNA levels before and after the outbreak of Zika virus | 6 months before the outbreak of Zika virus ; 12 months of the outbreak of Zika virus; First 6 months after the outbreak of Zika virus
  All biological results for HIV1 RNA will be collected retrospectivelly : 6 months before the outbreak of Zika virus , 12 months of the outbreak of Zika virus and 6 months after the outbreak of Zika virus in order to observe its evolution

CONTACTS AND LOCATIONS:
Overall Officials: Andre CABIE, MD, Principal Investigator — University Hospital of Martinique; Bruno HOEN, MD, Principal Investigator — University Hospital of Gaudeloupe; Andre CABIE, MD, Study Director — University Hospital of Martinique
Locations (2):
- University Hospital of Guadeloupe, Pointe-à-Pitre, Guadeloupe
- University Hospital of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No